CLINICAL TRIAL: NCT03849885
Title: Cutibacterium Dermal Colonization: Implications for Total Hip Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Colorado Joint Replacement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1378012
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Degenerative Osteoarthritis
MeSH Terms: conditions — Joint Diseases | interventions — clindamycin phosphate benzoyl peroxide combination; Benzoyl Peroxide

STUDY DESIGN:
Intervention Model Description: Group 1 - 4 %Chlorohexidine Wipe Group 2 - 4 % Chlorohexidine Wipe with 5% benzoyl peroxide (BPO) application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Skin Prep (No Intervention): Patients will undergo a skin cleansing protocols using 4% Chlorhexidine gluconate (CHG) cloths.
  After the skin prep, three 3-mm punch (Acu-Punch, Acuderm, Fort Lauderdale, FL) skin biopsies will performed for both an anterior-based hypothetical incision, and for a more lateral/posterior incision, for a total of 6 biopsies taken per subject.
- Experimental Skin Prep with BPO (Experimental): Patients will undergo a skin cleansing protocols using 4% Chlorhexidine gluconate (CHG) cloths.
  Following the CHG wipes, patients will be prepped with 5% BPO gel applied directly to the biopsy site.
  After the skin prep, three 3-mm punch (Acu-Punch, Acuderm, Fort Lauderdale, FL) skin biopsies will performed for both an anterior-based hypothetical incision, and for a more lateral/posterior incision, for a total of 6 biopsies taken per subject.
  Interventions: Drug: Benzoyl peroxide gel

INTERVENTIONS:
Drug: Benzoyl peroxide gel — Skin prep with Chlorohexidine wipes and BPO.
  Other Names: Acne Medication
  Arms: Experimental Skin Prep with BPO

SUMMARY:
This study is being done to investigate the colonization rate(growth rate) of a particular type of low-virulence (does not typically cause infection) bacterium called Propionibacterium, more specifically P acnes, the same bacterium that is responsible for the majority of acne. Information affecting hip surgery is currently unknown.

DETAILED DESCRIPTION:
This study is being done to investigate the colonization rate(growth rate) of a particular type of low-virulence (does not typically cause infection) bacterium called Propionibacterium. The most common bacterium of this family is P acnes, the same bacterium that is responsible for the majority of acne. There is increasing evidence that infection with P acnes and other Propionibacterium is a significant source of failure following certain orthopaedic shoulder procedures. However, information affecting hip surgery is currently unknown. Our personal experience leads us to believe that the numbers are actually quite high, since we are seeing an increased rate of Propionibacterium infection of hip replacement in the community. However, this type of study has never been done before, and therefore we simply do not know an accurate estimate for the average hip replacement patient's risk for Propionibacterium infection following hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 to 79 85 years of age
* CJR primary joint arthroplasty patients who are receiving care at Porter Adventist Hospital
* CJR established primary knee or hip arthroplasty patients with a native hip joint (no replacement on the biopsy side) who volunteers as a research participant.
* CJR patients without a previous arthroplasty procedure who have established care with our practice.

Exclusion Criteria:

* Previous history of hip infection
* Current antibiotic use or antibiotic use within the past week
* Previous history of Cutibacterium joint infection
* Current immunodeficiency disease or disorder
* Patients with active psoriatic disease or other focal inflammation over the hip
* Previous total hip arthroplasty (bilateral for the case of TKA patients and healthy volunteers, contralateral for THA patients)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Propionibacterium colinization rate on hips of healthy subjects | Tissues samples taken at the time of surgery will be held for 14 days
  The rate at which Propionibacterium could be isolated from the skin of healthy subjects at locations corresponding to both the direct anterior and posterior surgical approaches with and without intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Jennings, MD DPT, Principal Investigator — Colorado Joint Replacement
Locations (1):
- Colorado Joint Replacement, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared

REFERENCES:
- [Background] Butler-Wu SM, Burns EM, Pottinger PS, Magaret AS, Rakeman JL, Matsen FA 3rd, Cookson BT. Optimization of periprosthetic culture for diagnosis of Propionibacterium acnes prosthetic joint infection. J Clin Microbiol. 2011 Jul;49(7):2490-5. doi: 10.1128/JCM.00450-11. Epub 2011 May 4. PMID 21543562
- [Background] Dizay HH, Lau DG, Nottage WM. Benzoyl peroxide and clindamycin topical skin preparation decreases Propionibacterium acnes colonization in shoulder arthroscopy. J Shoulder Elbow Surg. 2017 Jul;26(7):1190-1195. doi: 10.1016/j.jse.2017.03.003. Epub 2017 May 4. PMID 28479255
- [Background] Heckmann N, Sivasundaram L, Heidari KS, Weber AE, Mayer EN, Omid R, Vangsness CT Jr, Hatch GF 3rd. Propionibacterium Acnes Persists Despite Various Skin Preparation Techniques. Arthroscopy. 2018 Jun;34(6):1786-1789. doi: 10.1016/j.arthro.2018.01.019. Epub 2018 Mar 24. PMID 29580742
- [Background] Heckmann N, Sivasundaram L, Lieberman JR. Propionibacterium acnes Infection in the Native Hip: A Case Report. JBJS Case Connect. 2015 Jul-Sep;5(3):e60. doi: 10.2106/JBJS.CC.N.00192. PMID 29252848
- [Background] Holinka J, Bauer L, Hirschl AM, Graninger W, Windhager R, Presterl E. Sonication cultures of explanted components as an add-on test to routinely conducted microbiological diagnostics improve pathogen detection. J Orthop Res. 2011 Apr;29(4):617-22. doi: 10.1002/jor.21286. Epub 2010 Dec 7. PMID 21337398
- [Background] Hsu JE, Neradilek MB, Russ SM, Matsen FA 3rd. Preoperative skin cultures are predictive of Propionibacterium load in deep cultures obtained at revision shoulder arthroplasty. J Shoulder Elbow Surg. 2018 May;27(5):765-770. doi: 10.1016/j.jse.2018.01.021. Epub 2018 Mar 12. PMID 29544667
- [Background] Hudek R, Sommer F, Kerwat M, Abdelkawi AF, Loos F, Gohlke F. Propionibacterium acnes in shoulder surgery: true infection, contamination, or commensal of the deep tissue? J Shoulder Elbow Surg. 2014 Dec;23(12):1763-1771. doi: 10.1016/j.jse.2014.05.024. Epub 2014 Aug 29. PMID 25179369
- [Background] Koh CK, Marsh JP, Drinkovic D, Walker CG, Poon PC. Propionibacterium acnes in primary shoulder arthroplasty: rates of colonization, patient risk factors, and efficacy of perioperative prophylaxis. J Shoulder Elbow Surg. 2016 May;25(5):846-52. doi: 10.1016/j.jse.2015.09.033. Epub 2015 Dec 15. PMID 26704361
- [Background] Kurtz SM, Lau E, Watson H, Schmier JK, Parvizi J. Economic burden of periprosthetic joint infection in the United States. J Arthroplasty. 2012 Sep;27(8 Suppl):61-5.e1. doi: 10.1016/j.arth.2012.02.022. Epub 2012 May 2. PMID 22554729
- [Background] Lavergne V, Malo M, Gaudelli C, Laprade M, Leduc S, Laflamme P, Rouleau DM. Clinical impact of positive Propionibacterium acnes cultures in orthopedic surgery. Orthop Traumatol Surg Res. 2017 Apr;103(2):307-314. doi: 10.1016/j.otsr.2016.12.005. Epub 2017 Jan 5. PMID 28065868
- [Background] Lee MJ, Pottinger PS, Butler-Wu S, Bumgarner RE, Russ SM, Matsen FA 3rd. Propionibacterium persists in the skin despite standard surgical preparation. J Bone Joint Surg Am. 2014 Sep 3;96(17):1447-50. doi: 10.2106/JBJS.M.01474. PMID 25187583
- [Background] Levy O, Iyer S, Atoun E, Peter N, Hous N, Cash D, Musa F, Narvani AA. Propionibacterium acnes: an underestimated etiology in the pathogenesis of osteoarthritis? J Shoulder Elbow Surg. 2013 Apr;22(4):505-11. doi: 10.1016/j.jse.2012.07.007. Epub 2012 Sep 13. PMID 22981447
- [Background] MacNiven I, Hsu JE, Neradilek MB, Matsen FA 3rd. Preoperative Skin-Surface Cultures Can Help to Predict the Presence of Propionibacterium in Shoulder Arthroplasty Wounds. JB JS Open Access. 2018 Feb 16;3(1):e0052. doi: 10.2106/JBJS.OA.17.00052. eCollection 2018 Mar 29. PMID 30229238
- [Background] Nelson CL, McLaren AC, McLaren SG, Johnson JW, Smeltzer MS. Is aseptic loosening truly aseptic? Clin Orthop Relat Res. 2005 Aug;(437):25-30. doi: 10.1097/01.blo.0000175715.68624.3d. PMID 16056022
- [Background] Ong KL, Kurtz SM, Lau E, Bozic KJ, Berry DJ, Parvizi J. Prosthetic joint infection risk after total hip arthroplasty in the Medicare population. J Arthroplasty. 2009 Sep;24(6 Suppl):105-9. doi: 10.1016/j.arth.2009.04.027. Epub 2009 Jun 2. PMID 19493644
- [Background] Parvizi J, Erkocak OF, Della Valle CJ. Culture-negative periprosthetic joint infection. J Bone Joint Surg Am. 2014 Mar 5;96(5):430-6. doi: 10.2106/JBJS.L.01793. PMID 24599206
- [Background] Phadnis J, Gordon D, Krishnan J, Bain GI. Frequent isolation of Propionibacterium acnes from the shoulder dermis despite skin preparation and prophylactic antibiotics. J Shoulder Elbow Surg. 2016 Feb;25(2):304-10. doi: 10.1016/j.jse.2015.08.002. Epub 2015 Oct 9. PMID 26456428
- [Background] Portillo ME, Corvec S, Borens O, Trampuz A. Propionibacterium acnes: an underestimated pathogen in implant-associated infections. Biomed Res Int. 2013;2013:804391. doi: 10.1155/2013/804391. Epub 2013 Nov 6. PMID 24308006
- [Background] Sabetta JR, Rana VP, Vadasdi KB, Greene RT, Cunningham JG, Miller SR, Sethi PM. Efficacy of topical benzoyl peroxide on the reduction of Propionibacterium acnes during shoulder surgery. J Shoulder Elbow Surg. 2015 Jul;24(7):995-1004. doi: 10.1016/j.jse.2015.04.003. PMID 26067191
- [Background] Scheer VM, Bergman Jungestrom M, Lerm M, Serrander L, Kalen A. Topical benzoyl peroxide application on the shoulder reduces Propionibacterium acnes: a randomized study. J Shoulder Elbow Surg. 2018 Jun;27(6):957-961. doi: 10.1016/j.jse.2018.02.038. Epub 2018 Mar 30. PMID 29609999
- [Background] Sierra JM, Garcia S, Martinez-Pastor JC, Tomas X, Gallart X, Vila J, Bori G, Macule F, Mensa J, Riba J, Soriano A. Relationship between the degree of osteolysis and cultures obtained by sonication of the prostheses in patients with aseptic loosening of a hip or knee arthroplasty. Arch Orthop Trauma Surg. 2011 Oct;131(10):1357-61. doi: 10.1007/s00402-011-1307-4. Epub 2011 May 11. PMID 21559986
- [Background] Wildeman P, Bruggemann H, Scholz CF, Leimbach A, Soderquist B. Propionibacterium avidum as an Etiological Agent of Prosthetic Hip Joint Infection. PLoS One. 2016 Jun 29;11(6):e0158164. doi: 10.1371/journal.pone.0158164. eCollection 2016. PMID 27355425
- [Background] Zeller V, Ghorbani A, Strady C, Leonard P, Mamoudy P, Desplaces N. Propionibacterium acnes: an agent of prosthetic joint infection and colonization. J Infect. 2007 Aug;55(2):119-24. doi: 10.1016/j.jinf.2007.02.006. Epub 2007 Apr 5. PMID 17418419
- [Background] Zeller VA, Letembet VA, Meyssonnier VA, Heym B, Ziza JM, Marmor SD. Cutibacterium (Formerly Propionibacterium) avidum: A Rare but Avid Agent of Prosthetic Hip Infection. J Arthroplasty. 2018 Jul;33(7):2246-2250. doi: 10.1016/j.arth.2018.02.008. Epub 2018 Feb 12. PMID 29544969